CLINICAL TRIAL: NCT02967913
Title: Urinary Symptoms and the Omission of the Bladder Flap at the Time of Primary Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Naval Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amy L O'Boyle, Staff Female Pelvic Medicine & Reconstructive Surgeon, National Naval Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2007.0005
Record Dates: First submitted 2016-11-07; First posted 2016-11-18 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Pelvic Floor Disorders
Keywords: Cesarean delivery; Obstetrical delivery; PFDI-20; UDI-6; Bladder flap
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bladder flap performed as per routine (Experimental): Bladder flap surgical step performed at time of non-urgent primary cesarean delivery as per routine
  Interventions: Procedure: Bladder flap
- Bladder flap is omitted (No Intervention): No bladder flap performed at time of non-urgent primary cesarean delivery

INTERVENTIONS:
Procedure: Bladder flap — bladder is separated from the lower uterine segment prior to making the uterine incision at time of cesarean delivery
  Other Names: Dissection of the vesicouterine fold
  Arms: Bladder flap performed as per routine

SUMMARY:
The bladder flap at the time of cesarean delivery is the term used to describe the separation of the bladder from the lower uterine segment by sharply incising the vesico-uterine peritoneum or serosa and using blunt and/or sharp dissection to develop this potential space which facilitates placement of a retractor, known as the bladder blade. Creating a bladder flap at the time of cesarean delivery is largely based on individual practice patterns and practitioners are divided in their use of this step. While creating a bladder flap has a theoretical advantage of protecting the bladder from injury, it is unknown whether this step has an effect on postoperative bladder function. The purpose of this study was to evaluate whether the omission or creation of a bladder flap results in a change in urinary symptoms as measured by the UDI-6 component of the PFDI-20.

DETAILED DESCRIPTION:
This is a Parallel Assignment design study. The PFDI-20 symptom questionnaire was completed upon enrollment. After the patient was prepped and draped, the operating room nurse opened a sealed opaque envelope marked with the study subject number containing a card marked with the assignment to bladder flap or no bladder flap, which was shown to the surgeons prior to the skin incision. The patient did not see the allocation nor was it verbalized in the operating room. The PFDI-20 was repeated 6-8 weeks after delivery at the patient's postpartum exam clinic visit. Equal number of bladder flap and no bladder flap assignment cards were randomly shuffled and placed in envelopes marked with the study subject ID number prior to the start of the study.

The study hypothesis was that the omission of the bladder flap at the time of primary cesarean delivery would be associated with lower urinary symptoms scores in the postpartum as measured by the UDI-6 component of the PFDI-20.

ELIGIBILITY:
Inclusion Criteria:

* pregnant at 37 weeks gestation or greater
* scheduled for a non-urgent primary cesarean delivery

Exclusion Criteria:

* pre-term (defined as less than 37 weeks 0 days gestation) prior pelvic surgery involving the bladder
* a diagnosis of any of the following conditions: endometriosis, uterine leiomyomata, chronic pelvic pain, urinary incontinence prior to pregnancy, nephrolithiasis during the current pregnancy,
* any circumstance that precluded adequate informed consent at the time of recruitment (such as a need to for urgent or emergent delivery)
* if the indication for cesarean was a failed trial of operative vaginal delivery (forceps or vacuum extraction)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The difference in urinary symptoms between study groups at 2 months postpartum | The difference in urinary symptoms between study groups at 2 months postpartum
  The difference in the urinary symptoms measured using the UDI-6 questionnaire at 2 months postpartum between study groups (bladder flap vs no bladder flap at time of primary cesarean delivery)

SECONDARY OUTCOMES:
Change in pelvic floor symptoms prior to delivery and at 2 months postpartum | During pregnancy and 2 months postpartum
  Change in the PFDI-20 and each sub scale before and after delivery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klein MC. Cesarean section on maternal request: a societal and professional failure and symptom of a much larger problem. Birth. 2012 Dec;39(4):305-10. doi: 10.1111/birt.12006. Epub 2012 Nov 5. PMID 23281950
- [Background] Rortveit G, Daltveit AK, Hannestad YS, Hunskaar S; Norwegian EPINCONT Study. Urinary incontinence after vaginal delivery or cesarean section. N Engl J Med. 2003 Mar 6;348(10):900-7. doi: 10.1056/NEJMoa021788. PMID 12621134
- [Background] Rortveit G, Hannestad YS, Daltveit AK, Hunskaar S. Age- and type-dependent effects of parity on urinary incontinence: the Norwegian EPINCONT study. Obstet Gynecol. 2001 Dec;98(6):1004-10. doi: 10.1016/s0029-7844(01)01566-6. PMID 11755545
- [Background] van Brummen HJ, Bruinse HW, van de Pol G, Heintz AP, van der Vaart CH. The effect of vaginal and cesarean delivery on lower urinary tract symptoms: what makes the difference? Int Urogynecol J Pelvic Floor Dysfunct. 2007 Feb;18(2):133-9. doi: 10.1007/s00192-006-0119-5. Epub 2006 Apr 21. PMID 16628375
- [Background] Wesnes SL, Lose G. Preventing urinary incontinence during pregnancy and postpartum: a review. Int Urogynecol J. 2013 Jun;24(6):889-99. doi: 10.1007/s00192-012-2017-3. Epub 2013 Feb 23. PMID 23436034
- [Background] Hohlagschwandtner M, Ruecklinger E, Husslein P, Joura EA. Is the formation of a bladder flap at cesarean necessary? A randomized trial. Obstet Gynecol. 2001 Dec;98(6):1089-92. doi: 10.1016/s0029-7844(01)01570-8. PMID 11755558
- [Background] Berghella V, Baxter JK, Chauhan SP. Evidence-based surgery for cesarean delivery. Am J Obstet Gynecol. 2005 Nov;193(5):1607-17. doi: 10.1016/j.ajog.2005.03.063. PMID 16260200
- [Background] Tuuli MG, Odibo AO, Fogertey P, Roehl K, Stamilio D, Macones GA. Utility of the bladder flap at cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2012 Apr;119(4):815-21. doi: 10.1097/AOG.0b013e31824c0e12. PMID 22395144
- [Background] Dahlke JD, Mendez-Figueroa H, Rouse DJ, Berghella V, Baxter JK, Chauhan SP. Evidence-based surgery for cesarean delivery: an updated systematic review. Am J Obstet Gynecol. 2013 Oct;209(4):294-306. doi: 10.1016/j.ajog.2013.02.043. Epub 2013 Mar 1. PMID 23467047
- [Background] Jozwik M, Jozwik M, Lotocki W, Mironczuk J. Dysuria due to bladder distortion after repeat cesarean section. Gynecol Obstet Invest. 1998;45(4):279-80. doi: 10.1159/000009985. PMID 9623798
- [Background] Tinelli A, Malvasi A, Vittori G. Laparoscopic treatment of post-cesarean section bladder flap hematoma: A feasible and safe approach. Minim Invasive Ther Allied Technol. 2009;18(6):356-60. doi: 10.3109/13645700903201357. PMID 19929298
- [Background] Handa VL, Blomquist JL, Knoepp LR, Hoskey KA, McDermott KC, Munoz A. Pelvic floor disorders 5-10 years after vaginal or cesarean childbirth. Obstet Gynecol. 2011 Oct;118(4):777-84. doi: 10.1097/AOG.0b013e3182267f2f. PMID 21897313
- [Background] Boyles SH, Li H, Mori T, Osterweil P, Guise JM. Effect of mode of delivery on the incidence of urinary incontinence in primiparous women. Obstet Gynecol. 2009 Jan;113(1):134-141. doi: 10.1097/AOG.0b013e318191bb37. PMID 19104369
- [Background] Blaivas JG, Panagopoulos G, Weiss JP, Somaroo C. Validation of the overactive bladder symptom score. J Urol. 2007 Aug;178(2):543-7; discussion 547. doi: 10.1016/j.juro.2007.03.133. Epub 2007 Jun 14. PMID 17570417